CLINICAL TRIAL: NCT00787644
Title: A Randomized, Placebo-Controlled Pilot Study of Pioglitazone for the Treatment of Moderate to Severe Asthma in Obese Asthmatics. (The GLITZ Asthma Study)
Brief Title: Pilot Study of Pioglitazone for the Treatment of Moderate to Severe Asthma in Obese Asthmatics (Glitz Asthma)
Acronym: GLITZ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: new safety concerns which emerged about pioglitazone during the trial
Sponsor: University of Vermont (Other)
Collaborators: American Lung Association (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anne Dixon, M.D., University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLITZ Asthma
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Asthma; Obesity
Keywords: Asthma; Adipose Tissue; Asthmatics; Pioglitazone; Actos; Obesity; Exacerbation; Fat; Overweight; Leptin; Adiponectin; Wheezing; Vermont; Pulmonary; Lung
MeSH Terms: conditions — Asthma; Obesity; Platelet Glycoprotein IV Deficiency; Overweight; Respiratory Sounds | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Pioglitazone
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone tablets; 30 mg/day for 2 weeks; then increased to 45 mg/day until week 12 (approximately 3 months)
  Arms: 1
Drug: Placebo — Matching placebo (inert tablet)
  Arms: 2

SUMMARY:
Asthmatics who are significantly overweight tend to have more severe symptoms, more flare ups, and are more likely to have poorly-controlled asthma when compared to other asthmatics.

Researchers believe this occurs because excess adipose tissue (fat) in the bosy can cause higher-than-normal levels of leptin and lower levels of adiponectin in the blood.

The researchers of this study are testing a medication called pioglitazone in overweight asthmatics because they believe it can help regulate leptin and adiponectin and that this may improve symptoms of asthma.

DETAILED DESCRIPTION:
Participants in this study will be randomly assigned (like the flip of a coin) to pioglitazone or placebo (an inactive pill). They will be given study medication to take every day for 12 weeks (3 months).

Participants will complete a number of asthma-related questionnaires and a variety of pulmonary function tests. Participants will undergo physical exams, an electrocardiogram, and blood sampling to measure leptin, adiponectin, markers of inflammation, blood cell counts, glucose levels, BNP hormone levels, and liver function.

To monitor participants throughout the study, follow-up visits will be done at 2, 6, and 12 weeks after starting study drug. At these visits many of the pulmonary function tests and questionnaires will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosed by a physician at least 1 year prior to study enrollment
* Poorly-controlled asthma at study enrollment
* Non smokers (stopped smoking at least 1 year ago) and limited lifetime history of smoking
* Body mass index 30-60
* Responds to methacholine challenge test with PC20 of <16 mg/ml
* On a stable dose of inhaled corticosteroid for at least 4 weeks prior to study entry
* FEV1 > 60% predicted
* Able to obtain weekly weights at home

Exclusion Criteria:

* Systemic steroids within the past 4 weeks
* Lung pathology other than asthma
* Other significant non-pulmonary co-morbidities such as: coronary artery disease, peripheral vascular disease, cerebrovascular disease, congestive heart failure with an ejection fraction <50%, liver disease or elevated liver enzymes at baseline, malignancy (excluding non-melanoma skin cancers), AIDS, renal failure with serum creatinine >3.0, or disorders requiring steroid treatment such as vasculitis, lupus, rheumatoid arthritis
* B-type natriuretic peptide (BNP) >400pg/ml
* Pregnant or lactating
* Currently taking a beta blocker, a CYP2C8 inhibitor or inducer such as gemfibrozil or rifampin, a TZD (thiazolidinedione), or allergic to TZD
* Taking antioxidants (if taking a multivitamin must be on a stable regimen prior to enrollment)
* Illicit drug use within the past year
* Current/active upper respiratory infection (if active URI, wait until asymptomatic for 1 week to enroll)
* Asthma exacerbation within the past 4 weeks (includes ER, urgent care, or hospital visits due to asthma resulting in an increase in asthma-related medications)
* Undergoing evaluation for sleep apnea, or plans to institute treatment for sleep apnea (patients on a stable treatment regimen for sleep apnea for the last 3 months will be allowed to participate)
* Clinically significant abnormalities present on screening 12-lead electrocardiogram
* Women of childbearing potential using oral contraceptives who are not willing to use a second method of contraception during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Dixon, MD, Principal Investigator — The Vermont Lung Center at the University of Vermont
Locations (1):
- The Vermont Lung Center at the University of Vermont, Colchester, Vermont, United States

REFERENCES:
- [Background] Hashimoto Y, Nakahara K. Improvement of asthma after administration of pioglitazone. Diabetes Care. 2002 Feb;25(2):401. doi: 10.2337/diacare.25.2.401. No abstract available. PMID 11815521
- [Background] Lee KS, Kim SR, Park SJ, Park HS, Min KH, Jin SM, Lee MK, Kim UH, Lee YC. Peroxisome proliferator activated receptor-gamma modulates reactive oxygen species generation and activation of nuclear factor-kappaB and hypoxia-inducible factor 1alpha in allergic airway disease of mice. J Allergy Clin Immunol. 2006 Jul;118(1):120-7. doi: 10.1016/j.jaci.2006.03.021. Epub 2006 May 19. PMID 16815147
- See also: Asthma informational website — http://www.nhlbi.nih.gov/health/dci/Diseases/Asthma/Asthma_WhatIs.html
- See also: Asthma informational website — http://www.ginasthma.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants did not qualify for randomization as they had a negative methacholine.
Groups:
- 1. Pioglitazone: Pioglitazone: Pioglitazone tablets; 30 mg/day for 2 weeks; then increased to 45 mg/day until week 12 (approximately 3 months)
- 2. Placebo: Placebo: Matching placebo (inert tablet)
Period: Overall Study
Arm/Group | 1. Pioglitazone | 2. Placebo
Started | 12 | 11
Completed | 10 | 9
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Pioglitazone | 2. Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23
PC20 [Median (Standard Deviation); unit: mg/ml] | 1.60 (5.91) | 1.99 (3.08) | 1.90 (3.08)

OUTCOME MEASURES:

1. Primary Outcome: PC20
Description: Airway reactivity will be measured with methacholine challenge testing following ATS guidelines.
  This is the concentration of methacholine that produces a 20% decrease in lung function (measured by forced expiratory volume in 1 second)
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: mg/ml
Arm/Group | 1. Pioglitazone | 2. Placebo
Number analyzed (Participants) | 10 | 9
mg/ml | 5.08 (7.42) | 2.37 (15.22)

ADVERSE EVENTS:
Arm/Group | 1. Pioglitazone | 2. Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No